CLINICAL TRIAL: NCT00689741
Title: A Double-blind, Placebo-controlled, Randomised Study of the Efficacy of an HPV-16/18 VLP Vaccine in the Prevention of HPV-16 and/or HPV-18 Cervical Infection in Healthy Adolescent and Young Adult Women in North America and Brazil.
Brief Title: Efficacy Study of HPV-16/18 Vaccine (GSK 580299) to Prevent HPV-16 and/or -18 Cervical Infection in Young Healthy Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 580299/001
Record Dates: First submitted 2008-05-30; First posted 2008-06-04 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Papillomavirus
Keywords: HPV; vaccine
MeSH Terms: conditions — Papillomavirus Infections | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Biological: Cervarix
- B (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: Cervarix — 3 doses of IM injection
  Arms: A
Biological: placebo — 3 doses of IM injection of Al(OH)3 placebo
  Other Names: Cervarix
  Arms: B

SUMMARY:
The purpose of this phase IIB MedImmune-sponsored study was to evaluate the efficacy of the HPV-16/18 VLP vaccine in the prevention of infection with HPV-16 and/or HPV-18 in adolescent and young adult women. A vaccine that prevents, or even reduces, the incidence of the common types of high-risk HPVs, particularly HPV-16 and HPV-18, could result in significant reduction in the incidence of cervical cancer and cancer-related mortality, as well as a reduction in the incidence of surgical procedures following abnormal Pap smears.

ELIGIBILITY:
Inclusion Criteria:

* Female between and including 15 and 25 years of age at the time of screening (must not have reached 26th birthday)
* Written informed consent obtained from the subject prior to enrolment (for subjects below the legal age of consent, written informed consent must also be obtained from a parent or legal guardian of the subject)
* Free of obvious health problems, as established by medical history and a directed physical examination
* No more than 6 lifetime sexual partners prior to enrolment
* Intact uterus
* Subject must be of non-childbearing potential, i.e., either surgically sterilised or, if of childbearing potential, she must be abstinent or must be using an effective method of birth control for 30 days prior to vaccination, have a negative urine pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series
* For subjects not enrolled in the HPV epidemiology study (999910/106) and for subjects completing the study (999910/106) >90 days prior to enrolment in the present study: agreement to complete both entrance and exit study questionnaires concerning general personal information, and sexual, contraceptive, reproductive and other gynaecological medical history
* For subjects previously enrolled in the HPV epidemiology study (and who completed the study and an entrance questionnaire) ≤ 90 days prior to enrolment in the present study: agreement to complete the exit questionnaire only.
* Normal cervical cytology (Pap smear) at screening, using the Cytyc ThinPrep® Pap Test. A normal Pap smear must also be adequate for interpretation, including the presence of endocervical cells; a Pap smear that is normal but inadequate for interpretation must be repeated as part of the protocol
* Seronegative for HPV-16 and HPV-18 antibody by ELISA at screening
* HPV DNA PCR negative for high-risk HPV types by PCR at screening. Genotyping will be specified using a reverse line probe assay specific for the detection of high-risk HPV types such as HPV-16, HPV-18 and HPV-16/18-related phylogenetic types

Exclusion Criteria:

* Pregnant or lactating female
* Female planning to become pregnant during the first eight months of the study (months 0-8)
* Abnormal vaginal discharge at the time of entry (once these subjects have received therapy to eradicate any discharge they will be eligible to participate in study)
* Previous administration of any components of the investigational vaccine
* Chronic administration (defined as more than 14 days) of immuno-suppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Administration of immunoglobulin and/or any blood products within the three months (90 days) preceding the first dose of study vaccine or planned administration during the study period
* Planned administration / administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of study vaccine. Administration of routine Meningococcal, Hepatitis A, Hepatitis B, Influenza, and Diphtheria/Tetanus vaccine up to 8 days before the first dose of study vaccine is allowed
* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period
* Receiving or expecting therapy for external or internal condylomata. Subjects with external condylomata not requiring therapy are eligible to participate in the study
* Genital herpes disease involving the cervix or characterized (on examination or by history) by extensive external lesions. Subjects with a history of recurrent genital herpes disease characterized by limited external lesions are eligible to participate in the study
* History of an abnormal cervical cytology (Pap smear) test (other than a single prior report of ASCUS with a subsequent normal report)
* Treatment for cervical disease by ablative therapy (cryotherapy or laser ablation) or excisional therapy (laser cone biopsy, loop excision, cold-knife conization)
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* A family history of congenital or hereditary immunodeficiency
* Major congenital defects or serious chronic illness
* History of any neurologic disorders or seizures, with the exception of a single febrile seizure during childhood
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests
* Acute disease at the time of enrolment.
* Oral temperature ≥99.5°F (≥37.5°C) / axillary temperature ≥99.5°F (37.5°C) / rectal temperature ≥100.4°F (≥38.0°C) / tympanic temperature on oral setting ≥99.5°F (37.5°C) / tympanic temperature on rectal setting ≥100.4°F (≥38.0°C)
* History of chronic alcohol consumption and/or intravenous drug abuse within the past 2 years
* Known or suspected allergy to any vaccine component
* Hepatomegaly, right upper quadrant abdominal pain or tenderness

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1113 (Actual)
Dates: Start 2001-01; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Cervical infection with HPV-16 and/or HPV-18 | Throughout the study

SECONDARY OUTCOMES:
Persistent cervical infection with HPV-16 and/or HPV-18 | Throughout the study
Cytologically confirmed or histopathologically confirmed LSIL, HSIL, squamous cell cancer, or adenocarcinoma concurrently associated with HPV-16 and/or HPV-18 cervical infection | Throughout the study
Determination of viral load for HPV-16 and HPV-18 (by PCR) for both self-obtained and Pap smear cervical samples | Throughout the study
Cervical infection with HPV-16, HPV-18 and/or HPV-16/18-related phylogenetic types | Throughout the study
Persistent cervical infection with HPV-16, HPV-18 and/or HPV-16/18-related phylogenetic types | Throughout the study
Cytologically confirmed or histopathologically confirmed LSIL, HSIL, squamous cell cancer, adenocarcinoma concurrently associated with cervical infection with HPV-16; HPV-18 and/or HPV-16/18-related phylogenetic types. | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] David MP, Van Herck K, Hardt K, Tibaldi F, Dubin G, Descamps D, Van Damme P. Long-term persistence of anti-HPV-16 and -18 antibodies induced by vaccination with the AS04-adjuvanted cervical cancer vaccine: modeling of sustained antibody responses. Gynecol Oncol. 2009 Dec;115(3 Suppl):S1-6. doi: 10.1016/j.ygyno.2009.01.011. Epub 2009 Feb 12. PMID 19217149
- [Background] David MP et al. Long-term persistence of detectable anti-HPV-16 and anti-HPV-18 antibodies induced by CervarixTM: modelling of sustained antibody responses. Abstract presented at the 26th Annual Meeting of the ESPID. Graz, Austria, 13-17 May 2008.
- [Background] David M-P et al. Modeling of long-term persistence of anti-HPV-16 and anti-HPV-18 antibodies induced by an AS04-adjuvanted cervical cancer vaccine. Abstract presented at the European Research Organization on Genital Infection and Neoplasia (EUROGIN) International Multidisciplinary Conference. Nice, France, 12-15 November 2008.
- [Background] Descamps D, Hardt K, Spiessens B, Izurieta P, Verstraeten T, Breuer T, Dubin G. Safety of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine for cervical cancer prevention: a pooled analysis of 11 clinical trials. Hum Vaccin. 2009 May;5(5):332-40. doi: 10.4161/hv.5.5.7211. Epub 2009 May 20. PMID 19221517
- [Background] Descamps D et al. Safety of human papillomavirus (HPV)-16/18 AS04 adjuvanted vaccine for cervical cancer prevention: integrated summary of 11 clinical trials. Abstract presented at the 26th Annual Meeting of the ESPID. Graz, Austria, 13-17 May 2008.
- [Background] Harper DM, Franco EL, Wheeler C, Ferris DG, Jenkins D, Schuind A, Zahaf T, Innis B, Naud P, De Carvalho NS, Roteli-Martins CM, Teixeira J, Blatter MM, Korn AP, Quint W, Dubin G; GlaxoSmithKline HPV Vaccine Study Group. Efficacy of a bivalent L1 virus-like particle vaccine in prevention of infection with human papillomavirus types 16 and 18 in young women: a randomised controlled trial. Lancet. 2004 Nov 13-19;364(9447):1757-65. doi: 10.1016/S0140-6736(04)17398-4. PMID 15541448
- [Background] Rombo L et al. Tolerability of HPV-16/18 AS04-adjuvanted cervical cancer vaccine. Abstract presented at the European Research Organization on Genital Infection and Neoplasia (EUROGIN) International Multidisciplinary Conference. Nice, France, 12-15 November 2008.
- [Background] Verstraeten T, Descamps D, David MP, Zahaf T, Hardt K, Izurieta P, Dubin G, Breuer T. Analysis of adverse events of potential autoimmune aetiology in a large integrated safety database of AS04 adjuvanted vaccines. Vaccine. 2008 Dec 2;26(51):6630-8. doi: 10.1016/j.vaccine.2008.09.049. PMID 18845199
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] El-Zein M, Ramanakumar AV, Naud P, Roteli-Martins CM, de Carvalho NS, Colares de Borba P, Teixeira JC, Moscicki AB, Harper DM, Tyring SK, Ramjattan B, Dubin G, Franco EL; HPV-007 Study Group. Determinants of Acquisition and Clearance of Human Papillomavirus Infection in Previously Unexposed Young Women. Sex Transm Dis. 2019 Oct;46(10):663-669. doi: 10.1097/OLQ.0000000000001053. PMID 31464859
- [Derived] Ramanakumar AV, Naud P, Roteli-Martins CM, de Carvalho NS, de Borba PC, Teixeira JC, Blatter M, Moscicki AB, Harper DM, Romanowski B, Tyring SK, Ramjattan B, Schuind A, Dubin G, Franco EL; HPV-007 Study Group. Incidence and duration of type-specific human papillomavirus infection in high-risk HPV-naive women: results from the control arm of a phase II HPV-16/18 vaccine trial. BMJ Open. 2016 Aug 26;6(8):e011371. doi: 10.1136/bmjopen-2016-011371. PMID 27566633
- [Derived] Naud PS, Roteli-Martins CM, De Carvalho NS, Teixeira JC, de Borba PC, Sanchez N, Zahaf T, Catteau G, Geeraerts B, Descamps D. Sustained efficacy, immunogenicity, and safety of the HPV-16/18 AS04-adjuvanted vaccine: final analysis of a long-term follow-up study up to 9.4 years post-vaccination. Hum Vaccin Immunother. 2014;10(8):2147-62. doi: 10.4161/hv.29532. PMID 25424918
- [Derived] Aregay M, Shkedy Z, Molenberghs G, David MP, Tibaldi F. Model-based estimates of long-term persistence of induced HPV antibodies: a flexible subject-specific approach. J Biopharm Stat. 2013;23(6):1228-48. doi: 10.1080/10543406.2013.834917. PMID 24138429
- [Derived] Moscicki AB, Wheeler CM, Romanowski B, Hedrick J, Gall S, Ferris D, Poncelet S, Zahaf T, Moris P, Geeraerts B, Descamps D, Schuind A. Immune responses elicited by a fourth dose of the HPV-16/18 AS04-adjuvanted vaccine in previously vaccinated adult women. Vaccine. 2012 Dec 17;31(1):234-41. doi: 10.1016/j.vaccine.2012.09.037. Epub 2012 Oct 11. PMID 23063422
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 580299/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 580299/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 580299/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 580299/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 580299/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 580299/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register